CLINICAL TRIAL: NCT06533787
Title: Impact of Echocardiography on Management of Critically Ill Neonates
Status: Recruiting | Type: Observational
Sponsor: Sahar Abozkaly Mahmoud (Other)
Responsible Party: Sponsor-Investigator, Sahar Abozkaly Mahmoud, Resident doctor of pediatrics at Sohag university hospital, Sohag University
Organization: Sohag University (Other)
Other Study IDs: Soh-Med-24-07-08MS
Record Dates: First submitted 2024-07-30; First posted 2024-08-01 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Critical Illness; Echocardiography; Neonatology
MeSH Terms: conditions — Critical Illness | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Hemodynamically unstable neonates
  Interventions: Device: Echocardiography
- Group 2: Hemodynamically stable neonates
  Interventions: Device: Echocardiography

INTERVENTIONS:
Device: Echocardiography — Functional echocardiography assessment

SUMMARY:
The goal of the study was to estimate the outcome (mortality and morbidity) among hemodynamically unstable neonates, as well as the time to return to hemodynamic stability following the use of ECHO in the management of hemodynamically unstable neonates.

DETAILED DESCRIPTION:
-All patients will be subjected to : Full clinical examination for manifestation or signs of hemodynamic instability and daily thereafter until discharge.

An echocardiographic assessment using Vivid T8 Pro ( GE MEDICAL SYSTEMS ( CHINA ) CO, LTD.) is done if manifestations of hemodynamic instability or shock appeared.

The imaging planes were identified by transducer location (subxiphoid, apical, parasternal, suprasternal notch, and right parasternal). The segmental approach was used to describe all of the major cardiovascular structures in sequence.

Suggested plan of management will be as the following:

1. Neonates with low LVO and impaired left ventricular contractility: dobutamine at a dose of 5-20 μg/kg/min was given, and if no improvement, volume expansion as a single intravenous infusion of 10-20 ml/kg of the crystalloid solution was given. If still no improvement, hydrocortisone at a dose of 1 mg/kg every 4 h was added. If improvement was not achieved, epinephrine was added at a dose of 0.05-2.6 μg/kg/min [11].
2. Neonates with LVO and hypovolemia (under-filled left ventricle): volume expansion as a single intravenous infusion of 10-20 ml/kg of the crystalloid solution will be given. If still no improvement, it was repeated [11].
3. Neonates with normal or high LVO without PDA: dopamine at a dose of 5-20 μg/kg/min is given. If no improvement, hydrocortisone at a dose of 1 mg/kg every 4 h is added. If improvement was not achieved, epinephrine is added at a dose of 0.05-2.6 μg/kg/min [11].
4. Neonates with normal or high LVO and hemodynamically significant PDA: PDA will be treated either medically or surgically [11].
5. During the current study period, all previously mentioned hemodynamically unstable neonate values were compared to values collected from the controlled group (200 hemodynamically stable neonates).
6. Neonates will be monitored regularly and subjected to repeated echocardiographic and clinical examinations to detect clinical and laboratory findings suggestive of hemodynamic instability or shock.

ELIGIBILITY:
Inclusion Criteria:

* All neonates ( age 0 to 28 days) admitted to the NICU of Sohag University Hospital during the period of the study in whom manifestations of hemodynamic instability or critical illness were elected regardless of gestational age, weight, gender, or type of disease.

Exclusion Criteria:

* Failure to obtain informed consent .
* Presence of congenital heart disease apart from PDA , PFO & small ASD .

Ages: 2 Hours to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Neonates ( age 0 to 28 days) admitted to the NICU of Sohag University Hospital during the period of the study
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Functional echocardiography ( ejection fraction using M mode echocardiography) | Repeat echocardiographic assessment on a daily basis ( 24 hours interval)
Functional echocardiography fraction shortening by M mode echocardiography | Repeat echocardiographic assessment on a daily basis ( 24 hours interval)
Assessment of ductus arteriosus ( diameter, shunt directionality ) by 2D and color doppler echocardiography | Repeat echocardiographic assessment 5 days after the first echo assessment
Assessment of pulmonary hypertension | Repeat echocardiographic assessment on a daily basis ( 24 hours interval) following proposed treatment of pulmonary hypertension
  Using peak tricuspid regurgitation velocity by colour doppler
Assessment of LV cardiac index | Repeat echocardiographic assessment on a daily basis ( 24 hours interval)
  Assessment of LV outflow tract diameter by 2D/M mode echocardiography in parasternal long axis view and assessment of Velocity-time integral of PW in LV outflow tract by PW doppler in apical five-chamber view
Assessment of RV cardiac index | Repeat echocardiographic assessment on a daily basis ( 24 hours interval)
  Assessment of RV outflow tract diameter by 2D echocardiography and Velocity-time integral of PW in RV outflow tract
Assessment of SVC flow | Repeat echocardiographic assessment on a daily basis ( 24 hours interval)
  Assessment of SVC diameter (mean of systolic and diastolic diameter) by M mode echocardiography in high parasternal view
Assessment of RV function | Repeat echocardiographic assessment on a daily basis ( 24 hours interval)
  Measurement of Tricuspid annular plane systolic excursion (TAPSE) using M mode echocardiography in apical four chamber view

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kluckow M, Seri I, Evans N. Functional echocardiography: an emerging clinical tool for the neonatologist. J Pediatr. 2007 Feb;150(2):125-30. doi: 10.1016/j.jpeds.2006.10.056. No abstract available. PMID 17236886
- [Background] Soleymani S, Borzage M, Seri I. Hemodynamic monitoring in neonates: advances and challenges. J Perinatol. 2010 Oct;30 Suppl:S38-45. doi: 10.1038/jp.2010.101. PMID 20877406
- [Background] Tibby SM, Hatherill M, Marsh MJ, Murdoch IA. Clinicians' abilities to estimate cardiac index in ventilated children and infants. Arch Dis Child. 1997 Dec;77(6):516-8. doi: 10.1136/adc.77.6.516. PMID 9496187
- [Background] Egan JR, Festa M, Cole AD, Nunn GR, Gillis J, Winlaw DS. Clinical assessment of cardiac performance in infants and children following cardiac surgery. Intensive Care Med. 2005 Apr;31(4):568-73. doi: 10.1007/s00134-005-2569-5. Epub 2005 Feb 15. PMID 15711976
- [Background] de Boode WP. Clinical monitoring of systemic hemodynamics in critically ill newborns. Early Hum Dev. 2010 Mar;86(3):137-41. doi: 10.1016/j.earlhumdev.2010.01.031. Epub 2010 Feb 20. PMID 20171815
- [Background] McNamara PJ, Sehgal A. Towards rational management of the patent ductus arteriosus: the need for disease staging. Arch Dis Child Fetal Neonatal Ed. 2007 Nov;92(6):F424-7. doi: 10.1136/adc.2007.118117. PMID 17951547
- [Background] Sehgal A, McNamara PJ. Does point-of-care functional echocardiography enhance cardiovascular care in the NICU? J Perinatol. 2008 Nov;28(11):729-35. doi: 10.1038/jp.2008.100. Epub 2008 Jul 17. PMID 18633423